CLINICAL TRIAL: NCT01311310
Title: Effect of Remote Ischemic Preconditioning on Children Undergoing Cardiac Surgery: Implication of Preoperative Cyanosis
Brief Title: Effect of Remote Ischemic Preconditioning on Children Undergoing Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: H-0907-028-286
Record Dates: First submitted 2009-09-20; First posted 2011-03-09 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2011-03

CONDITIONS: Cyanosis
Keywords: troponin, open heart surgery, children
MeSH Terms: conditions — Cyanosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- remote ischemic preconditioning (Experimental)
  Interventions: Other: RIPC (remote ischemic preconditioning)

INTERVENTIONS:
Other: RIPC (remote ischemic preconditioning) — RIPC will be performed by four 5-min cycles of lower limb ischemia and 5 in reperfusion using blood-pressure cuff inflated to a pressure 15 mmHg greater than the systolic arterial pressure measured via arterial line.

SUMMARY:
This study is conducted in order to evaluate the effect of remote ischemic preconditioning on children undergoing cardiac surgery, especially focusing on possible differences according to preoperative cyanosis.

ELIGIBILITY:
Inclusion Criteria:

* open heart surgery under cardiopulmonary bypass: ventricular septal defect, tetralogy of Fallot

Exclusion Criteria:

* chromosomal defect
* airway and parenchymal lung disease blood disorder
* isolated atrail septal defect
* immunodeficiency

Ages: 1 Month to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2009-10; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
troponin level | within the 1 day after operation
  troponin level will be checked 1, 6, 12 and 24 hours after operation. Ater making a graph (troponin-time), area under the curve will bw calculated.

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul National University Hospital, Seoul, Seoul
  - Seoul national university hospital, Seoul